CLINICAL TRIAL: NCT04285281
Title: Oral Gabapentin and Median Nerve Neural Mobilization Versus Control in the Treatment of Carpal Tunnel Syndrome
Brief Title: Oral Gabapentin and Median Nerve Mobilization in the Treatment of Carpal Tunnel Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Francisco Unda Solano, Biomedicine Doctorate Program Investigator, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: CE0072015-02-03
Record Dates: First submitted 2020-02-23; First posted 2020-02-26 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Gabapentin; Pain management; Physiotherapy
MeSH Terms: conditions — Carpal Tunnel Syndrome; Agnosia | interventions — Gabapentin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gabapentin (Active Comparator): Participants will be treated with a maximum of 600 mg per day, subdivided in 2 intakes of 300 mg oral capsules each 12 hours during a time lapse of 4 weeks.
  Interventions: Drug: Gabapentin oral capsules
- Control group (No Intervention): Participants that belong to the no intervention arm will be assigned to a waiting list to receive treatment. The participants will not receive treatment for carpal tunnel syndrome during a time lapse of 4 weeks. After this period of time, participants will begin the best treatment available.
- Median nerve neural mobilization (Experimental): Non pharmaceutical, non invasive, physiotherapy technique; which consists of a passive and repetitive upper limb movement that seeks to induced median nerve gliding and incursions against surrounding connective tissue. Subjects will be treated 5 days per week during a total time lapse of 4 weeks.
  Interventions: Other: Median nerve neural mobilization

INTERVENTIONS:
Drug: Gabapentin oral capsules — Oral capsule pharmaceutical treatment.
  Other Names: Neurontin
  Arms: Gabapentin
Other: Median nerve neural mobilization — Manual therapy maneuver performed in the upper limb.
  Arms: Median nerve neural mobilization

SUMMARY:
The present randomized clinical trial will perform a comparison of the pain reduction effects produced by the application of a non invasive and non pharmacological median nerve neural mobilization (physiotherapy treatment), to those effects produced by Gabapentin and the absence of treatment, in subjects who suffer the signs and symptoms of carpal tunnel syndrome.

DETAILED DESCRIPTION:
The present randomized clinical trial will perform a comparison of the pain reduction effects produced by the application of a non invasive and non pharmacological median nerve neural mobilization (physiotherapy treatment), to those effects produced by Gabapentin and the absence of treatment, in subjects who suffer the signs and symptoms of carpal tunnel syndrome. Additionally, effects over the functionality of the affected upper limb will be evaluated and compared. Subjects will be invited to participate and randomly allocated to 3 different groups.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be medically diagnosed with unilateral carpal tunnel syndrome (with confirmative electrodiagnostic findings).
* Full understanding of written and spoken Spanish (language).
* Participants must freely consent to participate.
* The presence of positive Phalen and Tinel sign.
* The presence of carpal tunnel syndrome signs and symptoms

Exclusion Criteria:

* The lack to meet inclusion criterions, the presence of cognitive impairment, tumors, cancer, recent (affected) upper limb surgery or trauma, pregnancy, metabolic neuropathy, obesity (body mass index over 30), participants who are not employed, deformities of the (affected) upper limb, recent skin injuries or infections (in the affected upper limb), autoimmune inflammatory conditions or flu type symptoms, allergy to gabapentin, and also: participants must not be (during the present investigation) under any type of pain reducing treatment (conservative, homeopathic, invasive or not invasive).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2020-04-01 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-08-10 (Actual)

PRIMARY OUTCOMES:
Distal upper limb pain | Changes from baseline (measured immediately before the application of the first treatment) and immediately after the application of the last treatment at 4 weeks.
  Assessed through the visual analog scale (VAS). The VAS is a psychometric response scale. It is a measurement instrument for subjective characteristics or attitudes that cannot be directly measured.The VAS is the most frequently used method to assess pain intensity. The scale will be displayed as a horizontal 10-cm line labelled at each end by descriptors such as 'no pain' (the minimum and best outcome possible) and 'worse pain ever' (maximum and worst outcome possible). The participant will mark the line to indicate pain severity and it is simply quantified by measuring the distance in centimeters from 0 (no pain) to the patient's marked rating.

SECONDARY OUTCOMES:
Upper limb function | Changes from baseline (measured immediately before the application of the first treatment), and at 40 minutes after the application of the last treatment.
  Assessed through the quick Quick Disabilities of the Arm, Shoulder and Hand questionary (QuickDASH), which is a shortened version of the 30-item Disabilities of the Arm, Shoulder and Hand (DASH) instrument.The instrument administered to the participants will be a self-report questionnaire, that will rate the difficulty and interference of daily life on a 5 point Likert scale. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability).
Work Status at baseline | Measured immediately before the application of the first treatment
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Do you currently work?"
Work Status post treatment | Measured immediatly after the application of the last treatment.
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Do you currently work?"
Change in Work Task (Job Type) | Measured immediatly after the application of the last treatment.
  This measure is performed through the employed participant (full-time or part-time) answering in a dichotomous manner (yes or no) the question: "Did you change your job type or task?"
Tampa Scale for Kinesiophobia-17 (TSK-17) | Changes from baseline (measured immediately before the application of the first treatment), and at 60 minutes after the application of the last treatment.
  The Tampa Scale for Kinesiophobia-17 (TSK-17) is a 17-item questionnaire designed to assess the fear of movement and re-injury (kinesiophobia). Items are rated on a 4-point Likert scale (ranging from "strongly disagree" to "strongly agree"), yielding a total score that reflects the severity of pain-related fear avoidance beliefs. The standard total score range for the Tampa Scale for Kinesiophobia (TSK-17) is 17 to 68. It is calculated by summing 17 items, each scored 1-4, with four items reverse-scored. Higher scores indicate greater fear of movement; a score $\ge 37$ suggests clinical kinesiophobia.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Unda, PhD, Principal Investigator — Confederación Gallega de Discapacidad
Locations (1):
- Ciudad Hospitalaria Enrique Tejera, Valencia, Carabobo, Venezuela

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hesami O, Haghighatzadeh M, Lima BS, Emadi N, Salehi S. The effectiveness of gabapentin and exercises in the treatment of carpal tunnel syndrome: a randomized clinical trial. J Exerc Rehabil. 2018 Dec 27;14(6):1067-1073. doi: 10.12965/jer.1836420.210. eCollection 2018 Dec. PMID 30656171
- [Background] Taverner D, Lisbona MP, Segales N, Docampo E, Calvet J, Castro S, Benito P. [Efficacy of gabapentin in the treatment of carpal tunnel syndrome]. Med Clin (Barc). 2008 Mar 22;130(10):371-3. doi: 10.1157/13117468. Spanish. PMID 18381028
- [Background] Dosenovic S, Jelicic Kadic A, Miljanovic M, Biocic M, Boric K, Cavar M, Markovina N, Vucic K, Puljak L. Interventions for Neuropathic Pain: An Overview of Systematic Reviews. Anesth Analg. 2017 Aug;125(2):643-652. doi: 10.1213/ANE.0000000000001998. PMID 28731977
- [Background] Erdemoglu AK. The efficacy and safety of gabapentin in carpal tunnel patients: open label trial. Neurol India. 2009 May-Jun;57(3):300-3. doi: 10.4103/0028-3886.53287. PMID 19587471
- [Background] Sanz DR, Solano FU, Lopez DL, Corbalan IS, Morales CR, Lobo CC. Effectiveness of median nerve neural mobilization versus oral ibuprofen treatment in subjects who suffer from cervicobrachial pain: a randomized clinical trial. Arch Med Sci. 2018 Jun;14(4):871-879. doi: 10.5114/aoms.2017.70328. Epub 2017 Sep 26. PMID 30002707
- [Background] Rodriguez-Sanz D, Calvo-Lobo C, Unda-Solano F, Sanz-Corbalan I, Romero-Morales C, Lopez-Lopez D. Cervical Lateral Glide Neural Mobilization Is Effective in Treating Cervicobrachial Pain: A Randomized Waiting List Controlled Clinical Trial. Pain Med. 2017 Dec 1;18(12):2492-2503. doi: 10.1093/pm/pnx011. PMID 28340157
- [Background] Eren Y, Yavasoglu NG, Comoglu SS. The relationship between QDASH scale and clinical, electrophysiological findings in carpal tunnel syndrome. Adv Clin Exp Med. 2018 Jan;27(1):71-75. doi: 10.17219/acem/67947. PMID 29521045
- [Background] Yucel H, Seyithanoglu H. Choosing the most efficacious scoring method for carpal tunnel syndrome. Acta Orthop Traumatol Turc. 2015;49(1):23-9. doi: 10.3944/AOTT.2015.13.0162. PMID 25803249